CLINICAL TRIAL: NCT05767814
Title: Role of Ultrasonographic and Tissue Biomarkers in Optimization of Psoriatic and Seronegative Rheumatoid Arthritis Patients Selection and Treatment Outcomes of Biologic Therapies.
Brief Title: Optimization of Psoriatic and Seronegative Rheumatoid Arthritis Patients Selection and Treatment Outcomes of Biologic Therapies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alivernini Stefano, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2784
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Psoriatic Arthritis; Rheumatoid Arthritis
Keywords: synovial tissue
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- PsO patients at risk of PsA development
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- naive to treatment PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- TNF-inhibitor resistant PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- IL-17-inhibitor resistant PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- TNF-inhibitor induced remission PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- IL-17-inhibitor induced remission PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- c-DMARDs resistant PsA
  Interventions: Other: Phenotyping of synovial immune and stromal cells
- c-DMARDs resistant RA
  Interventions: Other: Phenotyping of synovial immune and stromal cells

INTERVENTIONS:
Other: Phenotyping of synovial immune and stromal cells — Generate a comprehensive cellular and molecular atlas of PsA by CITE-Seq (single cell protein and transcriptomics) and spatial transcriptomics of synovium of PsO at risk of developing PsA and PsA patients across different disease stages.

SUMMARY:
Different classes of biological targeted therapies (b-DMARDs) are available for psoriatic arthritis (PsA) and seronegative rheumatoid arthritis (RA) (TNF inhibitors, anti-IL23, anti-IL17). A variable percentage of subjects, however, does not respond the first b-DMARD. Musculoskeletal ultrasound (US) and synovial tissue analysis could provide useful information on the top of clinical variables to predict response. The primary aim of this project is to create a global single-cell RNA sequencing atlas of PsA synovitis and to evaluate the predictive value of clinical, US and synovial variables (inflammatory cells and synovial tissue-single cell signature) on disease trajectory outcome and treatment response.

Patients with PsA or seronegative RA at different disease stages will be enrolled. Clinical and US examination will be performed at baseline, 3, 6 and 12 months, while synovial biopsy at baseline and 6 months. The optimal combination of clinical, US and synovial variables to stratify treatment response will be developed. The sensitivity to change of US and synovial variables and their evaluation in patients achieving clinical remission will also be considered as secondary aims.

The expected results will help the optimisation of treatment strategies in patients with PsA and seronegative RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the CASPAR classification Criteria for PsA
* Patients fulfilling the 2010 ACR/EULAR classification criteria for RA
* Clinically active arthritis, with at least one joint clinically involved;
* Subject eligible to treatment (c-or b-DMARD) as indicated by the treating rheumatologist according to usual clinical practice
* Subjects with PsA in sustained clinical and ultrasound remission (MDA)
* Patients with PsO and arthralgia

Exclusion Criteria:

* Severe and uncontrolled infections such as sepsis and opportunistic infections.
* Patients who are currently included in any interventional clinical trial in PsA or RA.
* Patients treated with more than one biologics.
* Subjects who are impaired, incapacitated, or incapable of completing study-related assessments
* Subjects with active vasculitis of a major organ system, with the exception of rheumatoid nodules.
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to RA or PsA and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
* Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.
* Subjects who currently abuse drugs or alcohol.
* Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
* Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
* Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
* Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
* Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. PsO with arthralgia (at risk of PsA)
  2. Naïve-to treatment active early PsA
  3. Established PsA with active disease: non-responders to TNFi
  4. Established PsA with active disease: non-responders to IL-17i
  5. PsA in remission induced by TNFi
  6. PsA in remission induced by IL-17i
  7. Established PsA with active disease: non-responders to cDMARDs
  8. Established RA with active disease: non-responders to cDMARDs
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Minimal Disease Activity status achievement | 6 months
  This outcome will be recorded for all study cohorts
PsA development (Fulfilment of the CASPAR criteria) | 12 months
  This outcome will be recorded only for PsO patient with arthralgia at risk of PsA development
Remission maintenance | 12 months
  This outcome will be recorded only for PsA patients in sustained remission

CONTACTS AND LOCATIONS:
Locations (2):
- Division of Rheumatology, Rome, Italy
- School of Immunity and Infection, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No